CLINICAL TRIAL: NCT03981224
Title: Additional Blood Test Enhances Diagnostic Sensitivity of Relapse Detection and Predicts Survivals in High-risk Nasopharyngeal Carcinoma Patients With Post-radiation Detectable Plasma EBV DNA
Brief Title: The Value of Post-radiation Detectable Plasma EBV DNA in High-risk Nasopharyngeal Carcinoma Patients
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, Jin-Ching Lin, Taichung Veterans General Hospital
Other Study IDs: CE12117-1
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Radiotherapy; Epstein-Barr virus
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma EBV DNA concentrations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- plasma EBV DNA detectable: the NPC patient received curative treatment and post-treatment plasma EBV DNA was detectable.
- plasma EBV DNA undetectable: the NPC patient received curative treatment and post-treatment plasma EBV DNA was undetectable.

SUMMARY:
An additional blood test at 2-3 months after RT is a valuable biomarker in predicting treatment outcome for NPC patients. Patients with persistently detectable EBV DNA during re-staging survey 2-3 months after RT should strengthen adjuvant therapy due to very high subsequent relapse rate and poor survivals.

DETAILED DESCRIPTION:
One week post-radiation therapy (RT) blood test showing persistently detectable EBV DNA is a very poor prognostic factor for nasopharyngeal carcinoma (NPC) patients. We hypothesize that additional EBV DNA confirmation test could enhance diagnostic sensitivity of relapse detection and predict survivals.

We screened 706 newly diagnosed NPC patients who finished curative RT with or without chemotherapy from March 2001 to December 2012. Additional EBV DNA blood test was performed at re-staging survey 2-3 months after RT. The association between treatment outcome (tumor relapse and patients' survival) and this additional blood test along with various clinical parameters were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* histologically-proven nasopharyngeal carcinoma without distant metastasis (M0) at initial presentation
* NPC patients who finished curative RT with or without chemotherapy

Exclusion Criteria:

* initial present M1 disease
* Secondary primary cancer diagnosed within 5 years
* performance status (WHO scale) less than 2

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: locally advanced NPC patients who finished curative RT with or without chemotherapy
Sampling Method: Probability Sample
Enrollment: 706 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

PRIMARY OUTCOMES:
relapse-free survival (RFS) | 5 years
  From the end of treatment to clinical or pathological proven disease relapse

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Overall survival was calculated from the day of enrollment until death or the last follow-up visit

OTHER OUTCOMES:
locoregional failure-free survival (LRFFS) | 5 years
  locoregional failure-free survival was calculated from the day of enrollment until locoregional failure or the last follow-up visit
distant metastasis failure-free survival (DMFFS) | 5 years
  distant metastasis failure-free survival was calculated from the day of enrollment until distant metastasis or the last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ching Lin, M.D.,PhD, Principal Investigator — Taichung Veterans General Hospital